CLINICAL TRIAL: NCT01127373
Title: Pilot Study of Multi-Beam Intensity-Modulated Radiation Therapy for Node-Positive Breast Cancer Patients Requiring Treatment of the Internal Mammary Lymph Nodes
Brief Title: Multi-Beam Intensity-Modulated Radiation Therapy for Node-Positive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-025
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: Breast; Radiation; Multi-Beam Intensity-Modulated Radiation; post mastectomy; post partial mastectomy; node-positive breast cancer; 10-025
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- radiation therapy via multi-beam IMRT (Experimental): This is a single-arm feasibility study of multi-beam IMRT with daily set-up verification in the treatment of women with node-positive breast cancer who will receive radiation to the breast/chest wall and regional lymph nodes, including the internal mammary lymph nodes.
  Interventions: Radiation: Multi-Beam Intensity-Modulated Radiation Therapy; Behavioral: BreastQ questionnaire-

INTERVENTIONS:
Radiation: Multi-Beam Intensity-Modulated Radiation Therapy — IMRT with multiple beams will be utilized to treat the breast or chest wall and axillary, supraclavicular and internal mammary lymph nodes. Treatment will be delivered once a day, 5 days a week for approximately 5 weeks. All missed radiation treatment visits will be made up. Daily set-up error will be checked prior to the delivery of every treatment.
Behavioral: BreastQ questionnaire- — MSKCC Department of Surgery. For patients who received a mastectomy with or without reconstruction, the questionnaire will be administered at baseline and 5-7 months after treatment.

SUMMARY:
This study is being performed to understand the safety of a new radiation treatment called "Multi-Beam Intensity Modulated Radiation Therapy" ( IMRT). Currently, the standard way of giving radiation is with "simplified" IMRT, which uses only 2 beams of radiation. "Multi-beam" IMRT works by using 6-12 small radiation beams to give a more "tailored" or "customized" radiation dose to the breast, chest wall, and the lymph nodes. At the same time, multi-beam IMRT may allow the dose to the heart, lungs, and nearby tissue to be lowered, especially when the internal mammary lymph nodes need to be targeted by radiation.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥18 years
* An invasive primary breast cancer of any histology arising from breast parenchyma
* Patient must be status post mastectomy or partial mastectomy with an assessment of axillary nodes via sentinel lymph node biopsy and/or axillary lymph node dissection
* Pathologic confirmation of metastatic disease in at least one regional lymph node. Regional lymph nodes are defined as the ipsilateral axillary lymph nodes, ipsilateral supraclavicular lymph nodes, and ipsilateral internal mammary lymph nodes. Thus, any T stage is allowed as long as the N stage is ≥1 and M stage is 0.
* Patient signed study-specific consent form.

Exclusion Criteria:

* Patients with distant metastasis.
* Patients who are pregnant or breastfeeding.
* Patients with psychiatric or addictive disorders that would preclude obtaining informed consent.
* Time between initial diagnosis of breast cancer and start of radiation therapy exceeds 13 months.
* Estimated life expectancy judged to be less than one year by patient's treating radiation oncologist.
* Prior radiation therapy to the ipsilateral or contralateral breast or thorax.
* Primary breast cancer is a lymphoma or sarcoma histology.
* Patients with a history of non-skin malignancy <5 years prior to the diagnosis of breast cancer.
* Patients requiring radiation to the bilateral breasts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Powell, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Follow Up Only), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Follow Up Only), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (Follow Up Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Follow Up Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre (Follow Up Only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Follow Up Only), Uniondale, New York

REFERENCES:
- [Derived] Ho AY, Ballangrud A, Li G, Gupta GP, McCormick B, Gewanter R, Gelblum D, Zinovoy M, Mueller B, Mychalczak B, Dutta P, Borofsky K, Parhar P, Reyngold M, Braunstein LZ, Chawla M, Krause K, Freeman N, Siu CT, Cost Z, Arnold BB, Zhang Z, Powell SN. Long-Term Pulmonary Outcomes of a Feasibility Study of Inverse-Planned, Multibeam Intensity Modulated Radiation Therapy in Node-Positive Breast Cancer Patients Receiving Regional Nodal Irradiation. Int J Radiat Oncol Biol Phys. 2019 Apr 1;103(5):1100-1108. doi: 10.1016/j.ijrobp.2018.11.045. Epub 2018 Nov 30. PMID 30508620
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Started | 116
Completed | 104
Not Completed | 12
Not completed — Not Treated | 3
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: 1 participant is male. A deviation to treat him per protocol was submitted and approved because using multi-beam radiation as part of the study was the best way to treat the study participant's breast cancer.
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
Age, Continuous [Median (Full Range); unit: years] | 50 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 109
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 79
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 116

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Receiving Adjuvant Radiation Therapy Via Multi-beam IMRT Using Daily 3D Position Verification
Description: The purpose of this pilot study is to assess the feasibility of utilizing multi-beam IMRT in the adjuvant treatment of the breast and regional lymph nodes of women with node-positive breast cancer requiring coverage of the internal mammary lymph nodes. A feasibility rate of at least 90% is required, ie, treatment can be successfully planned and delivered for at least 90% of the patients.
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
Participants
  Discontinued IMRT due to disease progression | 1
  Completed IMRT | 111
  Ineligible | 4

2. Secondary Outcome: Number of Participants Evaluated for Acute and Late Cutaneous Toxicity
Description: Toxicity evaluated by utilizing the CTCAE version 3.0 grading system.
Time Frame: 5-7 months following the completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
Participants | 116

3. Secondary Outcome: Number of Participants Evaluated for Late Subcutaneous Fibrosis
Description: The radiation oncologist will score late subcutaneous fibrosis at 5-7 months following CoT, utilizing the CTCAE version 3.0 grading system.
Time Frame: 5-7 months following the completion of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
Participants
  Experienced Skin & subcutaneous tissue disorders | 1
  Did not experience skin & subcutaneous tissue diso | 115

4. Secondary Outcome: Mean FEV1 at Baseline
Description: Participants FEV1 (forced expiratory volume in 1 second) measured at baseline
Time Frame: Baseline
Measure: Mean (Full Range); unit: liters
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
liters | 2.6 [1.2 to 3.9]

5. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by FEV1/FVC (Forced Vital Capacity) (%)
Description: Severity of radiation pneumonitis (RP) measured by FEV1 Z (forced expiratory volume in 1 second) and FVC Z (forced vital capacity) for participants at baseline
Time Frame: Baseline
Measure: Mean (Full Range); unit: FEV1 / FVC percentage
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
FEV1 / FVC percentage | 80.1 [57 to 93]

6. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by DLCO/Diffuse Capacity of Lung for CO2(mL/Min/mmHg)
Description: Participant Pulmonary Function Test/PFTs and mean Community-Acquired Pneumonia/CAP scores will be taken at baseline and again at 6 months post radiation therapy
Time Frame: Baseline
Measure: Mean (Full Range); unit: mL/min/mmHg
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
mL/min/mmHg | 18.5 [10 to 30]

7. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by the Mean of Total Community-Acquired Pneumonia (CAP) Score
Description: Mean Community-Acquired Pneumonia/CAP scores will be taken at baseline and again at 6 months post radiation therapy. The questionnaire focuses on the presence of dyspnea, severity of dyspnea, presence of cough, and general health and generates a "CAP score." Low values indicate more severe symptoms. Means will be taken of total scores, from 1-100.
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
units on a scale | 84.8 [33.8 to 100]

8. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by FEV1/FVC (Forced Vital Capacity) (%)
Description: as for outcome 6
Time Frame: 6 months post radiation therapy
Measure: Mean (Full Range); unit: 1 sec/FEV1 (Liters)
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
1 sec/FEV1 (Liters) | 2.6 [1.0 to 3.69]

9. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by FEV1/FVC (Forced Vital Capacity) (%)
Description: Severity of radiation pneumonitis (RP) measured by FEV1 Z (forced expiratory volume in 1 second) and FVC Z (forced vital capacity) for participants 6 months from baseline.
Time Frame: 6 months post radiation therapy
Measure: Mean (Full Range); unit: FEV1 / FVC percentage
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
FEV1 / FVC percentage | 79.6 [64 to 98]

10. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by DLCO/Diffuse Capacity of Lung for CO2(mL/Min/mmHg)
Description: as for outcome 6
Time Frame: 6 months post radiation therapy
Measure: Mean (Full Range); unit: mL/min/mmHg
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
mL/min/mmHg | 18.8 [5 to 65]

11. Secondary Outcome: Severity of Radiation Pneumonitis (RP) Measured by the Mean of Total Community-Acquired Pneumonia (CAP) Score
Description: Mean Community-Acquired Pneumonia/CAP scores will be taken at 6 months post radiation therapy. The questionnaire focuses on the presence of dyspnea, severity of dyspnea, presence of cough, and general health and generates a "CAP score." Low values indicate more severe symptoms. Means will be taken of total scores, from 1-100.
Time Frame: 6 months post radiation therapy
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
units on a scale | 83.2 [34.4 to 100]

12. Secondary Outcome: Median Follow-up Period
Description: Median follow-up period of the enrolled cohort
Time Frame: up to 82 months post-radiation therapy
Measure: Median (Full Range); unit: months
Arm/Group | Radiation Therapy Via Multi-beam IMRT
Number analyzed (Participants) | 116
months | 53.4 [0 to 82]

ADVERSE EVENTS:
Time Frame: 5-7 months following the completion of radiation therapy, up to 82 months
Arm/Group | Radiation Therapy Via Multi-beam IMRT
All-Cause Mortality (participants affected / at risk) | 33/116
Serious Adverse Events (participants affected / at risk) | 10/116
Other Adverse Events (participants affected / at risk) | 3/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Via Multi-beam IMRT (N=116)
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Breast Infection (Infections and infestations) | 1
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 1
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Skin and subcutaneous tissue disorders) | 2
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Pain - Chest/thorax NOS (General disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Seizure (Nervous system disorders) | 2
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy Via Multi-beam IMRT (N=116)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis assoc w/ rad- (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT01127373/Prot_SAP_000.pdf